CLINICAL TRIAL: NCT01600742
Title: Vorinostat and Concomitant Whole Brain Radiation Therapy in Patients With Brain Metastases: A Randomized, Double-blind, Placebo-controlled, Phase II Study
Brief Title: Vorinostat and Concurrent Whole Brain Radiotherapy for Brain Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stops to provide the study drug.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201110052MB
Record Dates: First submitted 2012-04-23; First posted 2012-05-17 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Brain Metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT, placebo (Active Comparator)
  Interventions: Drug: Placebo
- WBRT and concurrent vorinostat (Experimental)
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Run-in phase:
  WBRT: 2.5 Gy per fraction per day, day 1 through day 5 every week for 15 days, to a total dose of 37.5Gy.
  Vorinostat: 400 mg/day during WBRT, day 1 through day 7 every week till one day after WBRT.
  Randomization phase:
  WBRT: 2.5 Gy per fraction per day, day 1 through day 5 every week for 15 days, to a total dose of 37.5Gy.
  Vorinostat or placebo: 400 or 300 mg/day during radiation therapy (based on the results of run-in phase), day 1 through day 7 every week till one day after WBRT.
  Arms: WBRT and concurrent vorinostat
Drug: Placebo — Randomization phase:
  WBRT: 2.5 Gy per fraction per day, day 1 through day 5 every week for 15 days, to a total dose of 37.5Gy.
  Vorinostat or placebo: 400 or 300 mg/day during radiation therapy (based on the results of run-in phase), day 1 through day 7 every week till one day after WBRT.
  Arms: WBRT, placebo

SUMMARY:
Vorinostat is a potent and well tolerated HDAC inhibitor. It has been reported to enhance radiosensitivity of cancer cells. We hypothesize that the addition of vorinostat to WBRT may increase therapeutic efficacy for patients with brain metastases.

DETAILED DESCRIPTION:
Whole brain radiotherapy (WBRT) is the treatment of choice for the majority of patients with brain metastases. Although WBRT yields high radiologic response rate (27~56%) and is effective in palliation of neurologic symptoms, the response duration is limited and neurologic progression remains the main cause of death in a significant number of patients.

Vorinostat is reasonably well tolerated and there is also compelling evidence that vorinostat may serve as a radiosensitizer. Preclinical studies of HDAC inhibition have also shown efficacy in neuron protection. These data suggest that the addition of vorinostat to the standard therapy of WBRT may potentially increase their therapeutic efficacy without increasing neurotoxicity, and support the rationale of this phase II trial of vorinostat with WBRT in patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of a malignancy (lung and breast cancers) and radiologic evidence of brain metastases that are not suitable for surgery or radiosurgery as judged on the basis of the lesion size, number, location and the patients' personal choices.
* Patients with controlled systemic disease for >6 weeks (as judged on a case by case situation)
* Age≧20 years
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≦3
* Life expectancy of ≧6 months
* No prior cranial radiotherapy
* Negative urine pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Measurable lesions by gadolinium-enhanced MRI or contrast-enhanced CT scans. (≧10mm on T1-weighted gadolinium enhanced MRI or contrast-enhanced CT)
* Patients must have adequate organ and marrow reserve measured within 7 days prior to randomization as defined below:

  1. Hemoglobin >8.0 gm/dL;
  2. Absolute neutrophil count > 1,000/mcL;
  3. Platelets >100,000/mcL;
  4. Total bilirubin ≤ 1.5 x UNL (upper normal limit);
  5. AST(SGOT)/ALT(SGPT) ≤ 2.5 x UNL; for patients with liver metastases, AST(SGOT)/ALT(SGPT) ≤ 5 x UNL is allowed;
  6. Serum creatinine ≤ 1.5 x UNL;
  7. PTT ≤ UNL;
  8. INR ≤ 1.5;
  9. Serum sodium, calcium, potassium, and magnesium levels are within normal limits.
* Patients (or a surrogate) must be able to comply with study procedures and sign informed consent.

Exclusion Criteria:

* Prior cranial RT.
* Known hypersensitivity to any of the components of vorinostat.
* Use of Valproic acid or other histone deacetylase inhibitor, ≤2 weeks prior to registration and during treatment.
* Uncontrolled infection.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the prescribed regimens or limit compliance with study requirements.
* History of myocardial infarction or unstable angina ≤6 months prior to registration or congestive heart failure (CHF) requiring use of ongoing maintenance therapy, or life-threatening ventricular arrhythmias.
* Inability to take oral medications.
* Receiving any other investigational agent.
* Congenital long QT syndrome.
* Prolonged QTc interval (>450 msec)
* Any of the following Category I drugs that are generally known to have a risk of causing Torsades de Pointes ≤7 days prior to registration: Quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine
* Any of the following:

  1. Pregnant women
  2. Nursing women
  3. Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the duration of the study and for 3 weeks after treatment has ended.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate brain-specific progression free survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
brain-specific PFS | from randomization to progression of brain metastasis or death, assessed up to 36 months
PFS | from randomization to progression or death, assessed up to 36 months
response rate | 6 months
time to neuro-cognitive progression | 12 months
time to neurologic progression | 12 months
HRQoL | 12 months
Overall survival | from randomization to death, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan